CLINICAL TRIAL: NCT06603558
Title: Post-marketing Surveillance Study to Evaluate the Safety and Effectiveness of Atogepant for the Prevention of Migraine in Korean Adult Patients
Brief Title: Post-Marketing Study to Assess the Safety and Effectiveness of Oral Atogepant in Korean Adult Participants for the Prevention of Chronic or Episodic Migraine
Acronym: Atogepant PMSS
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-480
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Migraine; Episodic Migraine; Migraine
Keywords: Chronic Migraine; Episodic Migraine; Migraine; Atogepant; Qulipta; Aquipta
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Atogepant: Participants will receive atogepant as prescribed by their physician according to the local label.
  Interventions: Drug: Atogepant

INTERVENTIONS:
Drug: Atogepant — Oral Tablet
  Other Names: Qulipta; Aquipta

SUMMARY:
Migraine is a neurological disease characterized by moderate or severe headache, associated with nausea, vomiting, and/or sensitivity to light and sound. The study will assess the safety and effectiveness of atogepant for the preventive treatment of migraine in Korean adult patients with chronic migraine or episodic migraine under routine clinical practice.

Atogepant is an approved drug for preventive treatment of migraine in adults. Approximately 3000 adult participants who are prescribed atogepant by their doctors will be enrolled in this study in Korea.

Participants will receive atogepant oral tablets as prescribed by their physician. Participants will be followed for up to week 12.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with migraine suitable for the treatment with atogepant according to the latest approved local label.
* Participants prescribed atogepant in accordance with the approved local label.

Exclusion Criteria:

* Participants with any contraindication to atogepant as listed on the latest approved local label.
* Participants currently participating in another clinical research except observational study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants who have been prescribed atogepant for preventive treatment migraine according to the latest approved local label in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of participants who reported serious adverse event (SAE)/drug reaction (SADR) | Up to approximately 16 Weeks
  Percentage (%) of participants who reported serious adverse event (SAE)/drug reaction (SADR)
Percentage (%) of participants who reported unexpected (not reflected in the latest approved label) adverse event (AE)/drug reaction (ADR) | Up to approximately 16 Weeks
  Percentage (%) of participants who reported unexpected (not reflected in the latest approved label) adverse event (AE)/drug reaction (ADR)
Percentage (%) of participants who reported known (labeled) ADR | Up to approximately 16 Weeks
  Percentage (%) of participants who reported known (labeled) ADR
Percentage (%) of participants who reported non-serious AE/ADR | Up to approximately 16 Weeks
  Percentage (%) of participants who reported non-serious AE/ADR
Percentage (%) of participants who reported the events related to important potential risks and missing information defined in the Risk Management Plan (RMP) | Up to approximately 16 Weeks
  Percentage (%) of participants who reported the events related to important potential risks and missing information defined in the RMP
Percentage (%) of participants with AE: overall summary | Up to approximately 16 Weeks
  Percentage (%) of participants with AE: overall summary
Percentage (%) of participants with common (>=5%) AE | Up to approximately 16 Weeks
  Percentage (%) of participants with common (>=5%) AE
Percentage (%) of participants with AE leading to treatment discontinuation | Up to approximately 16 Weeks
  Percentage (%) of participants with AE leading to treatment discontinuation
Percentage (%) of participants who reported treatment-related AE per the investigator causality assessment | Up to approximately 16 Weeks
  Percentage (%) of participants who reported treatment-related AE per the investigator causality assessment
Percentage (%) of participants who reported treatment-related serious AE per the investigator causality assessment | Up to approximately 16 Weeks
  Percentage (%) of participants who reported treatment-related serious AE per the investigator causality assessment

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- South Korea (4):
  - Hallym University Dongtan Sacred Heart Hospital /ID# 273581, Hwaseong, Gyeonggido
  - Seoul National University Hospital /ID# 271892, Seoul, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 271893, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 272639, Seoul, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-480